CLINICAL TRIAL: NCT05167266
Title: Immediate and Long Term Cognitive Improvement After Cognitive Versus Emotion Management Psychoeducation Programs: a Randomised Trial in Covid Patients With Neuropsychological Difficulties
Brief Title: Long-Covid: Treatment of Cognitive Difficulties
Acronym: COV-COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Fabienne COLLETTE, Research Director, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCOV21-1303
Record Dates: First submitted 2021-12-21; First posted 2021-12-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Cognitive Dysfunction
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive psychoeducation (Experimental): 1) The cognitive intervention is a 4-session, psycho-educative, integrative and multidimensional intervention designed to prevent post-acute cognitive symptoms. Each individual session will last 90' and will concern a specific cognitive domain:
  * Cognition in covid, fatigue and sleep
  * Working memory and attentional functioning
  * Executive functioning
  * Memory functioning
  The structure of the sessions will be similar: (1) explanation about (dys)functioning of processes associated to the domain of interest: (2) identification of problems in daily life translated into functional objectives (e.g. keeping papers organized; scheduling activities to avoid fatigue); (3) discovery and application of (meta)cognitive strategies.
  Material (videos, tips,…) will be provided that the patients can consult when needed. The patients will have a diary to complete to explain when they applied the content of the intervention in daily life, and how successful it was.
  Interventions: Behavioral: Psychoeducation
- Affective psychoeducation (Active Comparator): 2) The affective intervention is also a psychoeducation program based on four sessions, in which different strategies and resources will be proposed to increase self-efficacy for emotion management:
  * Recognizing emotions and affective states
  * Accepting and communicating emotions and difficulties
  * Accepting the uncertainty associated with difficulties
  * Behavioural activation
  Material (videos, tips,…) will be provided that the patients can consult when needed. The patients will have a diary to complete to explain when they applied the content of the intervention in daily life, and how successful it was.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — Psychoeducation refers to the process of providing education and information to those seeking or receiving mental health services.

SUMMARY:
The purpose of the study is to explore the potential effectiveness of two common low-dose interventions, one targeting cognitive difficulties and the other targeting affective difficulties on quality of life and cognition in people suffering from long-COVID with cognitive complaints.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to understand the information and consent forms;
* Medically stable and at least 3 months after positive PCR for Covid-19;
* Self-reported sufficiently good physical condition to attend the appointment;
* No major hearing or vision disorders;
* Cognitive complaints that place the person in the top 20% of dissatisfied functioning on the BRIEF or MMQ questionnaires;
* Poor objective performance supported by a score below the 20th percentile on one task of the cognitive battery.

Exclusion Criteria:

* Any chronic or remote neurological disorder (i.e. stroke, head trauma, epilepsy, tumor);
* Cognitive impairment (minor or major neurocognitive disorder; intellectual disability) preexisting to the Covid-19 episode;
* Acute brain injury or acute encephalopathy from another aetiology than covid (e.g., sepsis, liver or renal failure, alcohol or drug withdrawal, drug toxicity);
* Documented preexisting history of psychiatric illness, including substance abuse; Open-heart cardiac surgery or cardiac arrest during the last 6 months;
* Current hospitalization;
* Current revalidation care with cognitive treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Comparison of change in subjective cognitive difficulties between the two intervention arms | Two months post-intervention
  Subjective report of difficulties experienced by patients in daily life: BRIEF (Behavioral Rating Inventory of Executive Function) and MMQ (Multifactorial Memory Questionnaire) questionnaires.
  The BRIEF summary index scales (Behavioral Regulation Index and Metacognition Index) and the scale reflecting overall functioning (Global Executive Composite) are expressed at t-scores (M=50, SD=10) ranging from 30 to 100. Higher scores indicates better outcome.
  There are three scales in the MMQ : Satisfaction Scale, Ability Scale and Strategy Scale. The individual score will range from 0 to 72, from 0 to 80 and from 0 to 76 respectively for each scale. Higher scores indicate better ratings.

SECONDARY OUTCOMES:
Comparison of change in subjective cognitive difficulties between the two intervention arms | Eight months post-intervention
  Subjective report of difficulties experienced by patients in daily life: scores from BRIEF and MMQ questionnaires
  The BRIEF summary index scales (Behavioral Regulation Index and Metacognition Index) and the scale reflecting overall functioning (Global Executive Composite) are expressed at t-scores (M=50, SD=10) ranging from 30 to 100. Higher scores indicates better outcome.
  There are three scales in the MMQ : Satisfaction Scale, Ability Scale and Strategy Scale. The individual score will range from 0 to 72, from 0 to 80 and from 0 to 76 respectively for each scale. Higher scores indicate better ratings.
Comparison of change in quality of life assessment between the two intervention arms | 2 and 8 months post-intervention
  Subjective report of quality of life experienced by patients in daily life: scores from ISQV (Inventaire Systématique de Qualité de Vie) and EQ-5D (from the EuroQol Group).
  Scores at ISQV range from 1 (smallest possible gap between 'desired situation' and 'current situation' ) to 100 (largest possible gap). Scores at the EQ-5D range from 5 (full health) to 25 (worst health).
Comparison of changes in cognitive performance between the two intervention arms | 2 and 8 months post-intervention
  Cognitive scores in the domains of attention, working memory, long term memory and executive functions, as well as global cognitive efficiency.

OTHER OUTCOMES:
Comparison of Work productivity and activity impairment between the two intervention arms | 2 and 8 months post-intervention
  Scores at the WPAI (Work Productivity and Activity Impairment) scale. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
Comparison of fatigue level between the two intervention arms | 2 and 8 months post-intervention
  Score at the M-FIS scale (Modified Fatigue Impact Scale). The individual score will range from 0 [no fatigue] to 84 [extreme fatigue]
Comparison of sleep quality between the two intervention arms | 2 and 8 months post-intervention
  Score at the PSQI (Pittsburgh Sleep Quality Inventory) scale. The individual score will range from 0 to 21. Higher score indicates lower sleep quality
Comparison of psychological distress between the two intervention arms | 2 and 8 months post-intervention
  Score at the OQ-45 (Outcome Questionnaire 45) scale. Scores range from 0 to 180, Higher scores indicate more severe psychological distress and functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Willems, PhD, Study Director — ULiège; Fabienne Collette, PhD, Principal Investigator — ULiège
Locations (5):
- Belgium (5):
  - ULB - CHU Erasme, Brussels
  - CHC Mont Légia, Liège
  - CHR Citadelle, Liège
  - ULiège - CHU, Liège
  - ULiège - CPLU, Liège

IPD SHARING:
Plan to Share IPD: Yes
Research data upon request after publication of the main results
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Cabello Fernandez C, Didone V, Lesoinne A, Slama H, Fery P, Rousseau AF, Moutschen M; COVCOG group; Collette F, Willems S. Cognitive and affective psychoeducation for Long COVID: a randomized controlled trial. Brain Commun. 2025 Nov 11;7(6):fcaf447. doi: 10.1093/braincomms/fcaf447. eCollection 2025. PMID 41277895
- [Derived] Cabello Fernandez C, Didone V, Slama H, Dupuis G, Fery P, Delrue G, Lesoinne A, Collette F, Willems S. Profiles of Individuals With Long COVID Reporting Persistent Cognitive Complaints. Arch Clin Neuropsychol. 2025 Nov 24;40(8):1455-1472. doi: 10.1093/arclin/acaf064. PMID 40645608
- [Derived] Willems S, Didone V, Cabello Fernandez C, Delrue G, Slama H, Fery P, Goin J, Della Libera C; COVCOG Group; Collette F. COVCOG: Immediate and long-term cognitive improvement after cognitive versus emotion management psychoeducation programs - a randomized trial in covid patients with neuropsychological difficulties. BMC Neurol. 2023 Aug 18;23(1):307. doi: 10.1186/s12883-023-03346-9. PMID 37596541